CLINICAL TRIAL: NCT03626662
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 890 in Subjects With Elevated Plasma Lipoprotein(a)
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Study of AMG 890 in Subjects With Elevated Plasma Lipoprotein(a)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 20170544
Record Dates: First submitted 2018-06-19; First posted 2018-08-13 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-12

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The subjects and the investigative site staff, except for the unblinded pharmacist, will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Single Ascending Dose Cohorts
  Interventions: Drug: Placebo
- AMG 890 (Experimental): Single Ascending Dose Cohorts
  Interventions: Drug: AMG 890

INTERVENTIONS:
Drug: AMG 890 — Ascending Single Doses of AMG 890
  Arms: AMG 890
Drug: Placebo — Calculated volume to match experimental drug.
  Arms: Placebo

SUMMARY:
This is a first-in-human, randomized, double-blind, placebo-controlled, single ascending dose study in subjects with elevated plasma Lipoprotein(a) [Lp(a)]. AMG 890 will be evaluated in approximately 80 subjects to assess safety, tolerability, pharmacokinetics and pharmacodynamic effects.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with ages between 18 and 70 years old, inclusive.
* Protocol-defined elevated plasma Lp(a) level.
* Body mass index (BMI) greater than or equal to 18 and less than or equal to 40 kg/m2, at screening.
* Women must be of non-reproductive potential.
* Other Inclusion criteria may apply

Exclusion Criteria:

* Currently receiving treatment in another investigational device or drug study.
* Women who are lactating/breastfeeding or who plan to breastfeed while on study or through 90 days after receiving the last dose of investigational product (for subjects who withdraw prior to end of study).
* History or evidence of a clinically significant disorder, condition or disease that would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.
* History or clinical evidence of bleeding diathesis or any coagulation disorder.
* History or clinical evidence of peripheral neuropathy.
* Other Exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (9):
- United States (7):
  - Orange County Research Center, Tustin, California
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - QPS Miami Research Associates, South Miami, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - New York University, New York, New York
  - Medpace Inc, Cincinnati, Ohio
- Australia (2):
  - Clinical Medical and Analytical eXellence CMAX, Adelaide, South Australia
  - Linear Clinical Research Limited, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Koren MJ, Moriarty PM, Baum SJ, Neutel J, Hernandez-Illas M, Weintraub HS, Florio M, Kassahun H, Melquist S, Varrieur T, Haldar SM, Sohn W, Wang H, Elliott-Davey M, Rock BM, Pei T, Homann O, Hellawell J, Watts GF. Preclinical development and phase 1 trial of a novel siRNA targeting lipoprotein(a). Nat Med. 2022 Jan;28(1):96-103. doi: 10.1038/s41591-021-01634-w. Epub 2022 Jan 13. PMID 35027752
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 8 research centers in the United States (US) and Australia between July 2018 and April 2023.
Pre-assignment Details: Participants were randomized in a 3:1 ratio to receive either Olpasiran or a volume-matched placebo via subcutaneous (SC) injection, across 9 single ascending dose cohorts.
Groups:
- Placebo: Participants with screening plasma Lipoprotein(a) (Lp[a]) >=70 nmol/L and <199 nmol/L received placebo matching Olpasiran as a single SC injection on Day 1 in cohorts 1-5. Participants with screening plasma Lp(a) >=200 nmol/L received placebo matching Olpasiran as a single SC injection on Day 1 in cohorts 6-9.
- Cohort 1: Olpasiran 3 mg: Participants with screening plasma Lp(a) >=70 nmol/L and <199 nmol/L received Olpasiran 3 mg as a single SC injection on Day 1.
- Cohort 2: Olpasiran 9 mg: Participants with screening plasma Lp(a) >=70 nmol/L and <199 nmol/L received Olpasiran 9 mg as a single SC injection on Day 1.
- Cohort 3: Olpasiran 30 mg: Participants with screening plasma Lp(a) >=70 nmol/L and <199 nmol/L received Olpasiran 30 mg as a single SC injection on Day 1.
- Cohort 4 Olpasiran: 75 mg: Participants with screening plasma Lp(a) >=70 nmol/L and <199 nmol/L received Olpasiran 75 mg as a single SC injection on Day 1.
- Cohort 5 Olpasiran: 225 mg: Participants with screening plasma Lp(a) >=70 nmol/L and <199 nmol/L received Olpasiran 225 mg as a single SC injection on Day 1.
- Cohort 6: Olpasiran 9 mg: Participants with screening plasma Lp(a) >= 200 nmol/L received Olpasiran 9 mg as a single SC injection on Day 1. Participants were required to be on a stable dose of statin for at least 6 weeks prior to enrollment.
- Cohort 7: Olpasiran 75 mg: Participants with screening plasma Lp(a) >= 200 nmol/L received Olpasiran 75 mg as a single SC injection on Day 1. Participants were required to be on a stable dose of statin for at least 6 weeks prior to enrollment.
- Cohort 8: Olpasiran 225 mg: Participants with screening plasma Lp(a) >= 200 nmol/L received Olpasiran 225 mg as a single SC injection on Day 1. Participants were required to be on a stable dose of statin for at least 6 weeks prior to enrollment.
- Cohort 9: Olpasiran 675 mg: Participants with screening plasma Lp(a) >= 200 nmol/L received Olpasiran 675 mg as a single SC injection on Day 1. Participants were required to be on a stable dose of statin for at least 6 weeks prior to enrollment.
Period: Overall Study
Arm/Group | Placebo | Cohort 1: Olpasiran 3 mg | Cohort 2: Olpasiran 9 mg | Cohort 3: Olpasiran 30 mg | Cohort 4 Olpasiran: 75 mg | Cohort 5 Olpasiran: 225 mg | Cohort 6: Olpasiran 9 mg | Cohort 7: Olpasiran 75 mg | Cohort 8: Olpasiran 225 mg | Cohort 9: Olpasiran 675 mg
Started | 20 | 6 | 6 | 6 | 6 | 6 | 9 | 9 | 5 | 6
Participants Who Received Placebo in Cohorts 1-5 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Participants Who Received Placebo in Cohorts 6-9 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 17 | 6 | 4 | 6 | 2 | 3 | 8 | 6 | 5 | 5
Not Completed | 3 | 0 | 2 | 0 | 4 | 3 | 1 | 3 | 0 | 1
Not completed — Withdrawal of Consent from Study | 2 | 0 | 0 | 0 | 4 | 3 | 0 | 0 | 0 | 1
Not completed — Decision by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set consisted of all participants who received at least 1 dose of Olpasiran or placebo.
Groups:
- Placebo: Participants with screening plasma Lp(a) >=70 nmol/L and <199 nmol/L received placebo matching Olpasiran as a single SC injection on Day 1 in cohorts 1-5. Participants with screening plasma Lp(a) >=200 nmol/L received placebo matching Olpasiran as a single SC injection on Day 1 in cohorts 6-9.
- Total: Total of all reporting groups
Arm/Group | Placebo | Cohort 1: Olpasiran 3 mg | Cohort 2: Olpasiran 9 mg | Cohort 3: Olpasiran 30 mg | Cohort 4 Olpasiran: 75 mg | Cohort 5 Olpasiran: 225 mg | Cohort 6: Olpasiran 9 mg | Cohort 7: Olpasiran 75 mg | Cohort 8: Olpasiran 225 mg | Cohort 9: Olpasiran 675 mg | Total
Number analyzed (Participants) | 20 | 6 | 6 | 6 | 6 | 6 | 9 | 9 | 5 | 6 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (8.8) | 42.7 (16.0) | 50.2 (7.6) | 34.5 (11.5) | 51.5 (13.4) | 40.8 (14.3) | 52.7 (10.8) | 52.8 (8.3) | 58.2 (4.3) | 47.7 (13.1) | 49.2 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 2 | 1 | 3 | 0 | 3 | 3 | 4 | 1 | 29
  Male | 11 | 3 | 4 | 5 | 3 | 6 | 6 | 6 | 1 | 5 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 6 | 6 | 4 | 1 | 2 | 2 | 3 | 0 | 0 | 32
  Not Hispanic or Latino | 12 | 0 | 0 | 2 | 5 | 4 | 7 | 6 | 5 | 6 | 47
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 4 | 0 | 1 | 3 | 1 | 1 | 0 | 0 | 1 | 14
  White | 16 | 2 | 6 | 5 | 3 | 5 | 7 | 9 | 5 | 5 | 63
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event was defined as any untoward medical occurrence in a clinical trial participant. A TEAE was defined as any event with onset after the administration of the first dose of investigational product and up to and including the end of treatment date, or end of trial for participants who discontinued the trial during the treatment period. Clinically significant changes in vital signs, electrocardiograms (ECGs), and safety laboratory analytes were included as TEAEs.
Time Frame: From first dose of trial until the end of trial; median (min, max) duration was 8.54 (0.23, 23.92) months
Population: The safety analysis set consisted of all participants who received at least 1 dose of Olpasiran or placebo.
Measure: Count of Participants; unit: Participants
Groups:
- Cohorts 1-5: Placebo: Participants with screening plasma Lp(a) >=70 nmol/L and <199 nmol/L received placebo matching Olpasiran as a single SC injection on Day 1 in cohorts 1 -5.
- Cohorts 6-9: Placebo: Participants with screening plasma Lp(a) >=200 nmol/L received placebo matching Olpasiran as a single SC injection on Day 1 in cohorts 6-9.
Arm/Group | Cohorts 1-5: Placebo | Cohort 1: Olpasiran 3 mg | Cohort 2: Olpasiran 9 mg | Cohort 3: Olpasiran 30 mg | Cohort 4 Olpasiran: 75 mg | Cohort 5 Olpasiran: 225 mg | Cohorts 6-9: Placebo | Cohort 6: Olpasiran 9 mg | Cohort 7: Olpasiran 75 mg | Cohort 8: Olpasiran 225 mg | Cohort 9: Olpasiran 675 mg
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 10 | 9 | 9 | 5 | 6
Participants | 5 | 3 | 3 | 5 | 1 | 0 | 7 | 6 | 3 | 4 | 4

2. Secondary Outcome: Maximum Observed Concentration (Cmax) of Olpasiran
Description: Blood samples were collected for measurement of serum concentrations of Olpasiran.
Time Frame: Cohorts 1-5:pre-dose, Days 1-4, 7, 15, 29, 57, 85 post-dose; Cohorts 6-7:pre-dose, Days 1, 2, 4, 7, 15 post-dose; Cohort 8:pre-dose, Days 1, 2, 4, 7, 15, 29, 57, 85, 113 post-dose; Cohort 9:pre-dose, Days 1, 2, 4, 7, 15, 29, 57, 85, 113, 155 post-dose
Population: The pharmacokinetic (PK) analysis set consisted of all Olpasiran dosed participants for whom at least one PK parameter was reliably estimated.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: Olpasiran 3 mg | Cohort 2: Olpasiran 9 mg | Cohort 3: Olpasiran 30 mg | Cohort 4 Olpasiran: 75 mg | Cohort 5 Olpasiran: 225 mg | Cohort 6: Olpasiran 9 mg | Cohort 7: Olpasiran 75 mg | Cohort 8: Olpasiran 225 mg | Cohort 9: Olpasiran 675 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 9 | 9 | 5 | 6
ng/mL | 11.7 (2.36) | 36.1 (19.7) | 74.9 (25) | 252 (153) | 421 (223) | 17.4 (7.48) | 111 (56.3) | 1390 (947) | 2620 (888)

3. Secondary Outcome: Time to Reach Cmax (Tmax) of Olpasiran
Description: Blood samples were collected for measurement of serum concentrations of Olpasiran.
Time Frame: as for outcome 2
Population: The PK analysis set consisted of all Olpasiran dosed participants for whom at least one PK parameter was reliably estimated.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1: Olpasiran 3 mg | Cohort 2: Olpasiran 9 mg | Cohort 3: Olpasiran 30 mg | Cohort 4 Olpasiran: 75 mg | Cohort 5 Olpasiran: 225 mg | Cohort 6: Olpasiran 9 mg | Cohort 7: Olpasiran 75 mg | Cohort 8: Olpasiran 225 mg | Cohort 9: Olpasiran 675 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 9 | 9 | 5 | 6
hours | 3.0 [1.0 to 9.0] | 3.0 [3.0 to 6.0] | 7.5 [1.0 to 9.0] | 4.5 [0.17 to 9.0] | 6.0 [1.0 to 12] | 3.0 [1.0 to 9.0] | 6.0 [3.0 to 24] | 3.0 [1.0 to 23] | 4.5 [2.1 to 6.2]

4. Secondary Outcome: Area Under the Concentration-time Curve (AUC) From Time Zero to the Last Quantifiable Timepoint (AUC0-last) of Olpasiran
Description: Blood samples were collected for measurement of serum concentrations of Olpasiran.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hour*ng/mL
Arm/Group | Cohort 1: Olpasiran 3 mg | Cohort 2: Olpasiran 9 mg | Cohort 3: Olpasiran 30 mg | Cohort 4 Olpasiran: 75 mg | Cohort 5 Olpasiran: 225 mg | Cohort 6: Olpasiran 9 mg | Cohort 7: Olpasiran 75 mg | Cohort 8: Olpasiran 225 mg | Cohort 9: Olpasiran 675 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 9 | 9 | 5 | 6
hour*ng/mL | 116 (39.8) | 352 (141) | 1020 (329) | 2830 (730) | 7800 (1670) | 240 (96.3) | 2060 (642) | 29600 (23500) | 44800 (16400)

5. Secondary Outcome: Change From Baseline in Plasma Lp(a) Levels
Description: Change from baseline for plasma Lp(a) by cohort and at scheduled time points were presented.
Time Frame: Cohorts 1-2:Baseline,Days 2,4,7,15,18,22,29,43,57,71,85,113;3-5:Baseline,Days 2,4,7,15,18,22,29,43,57,71,85,113,155,183,225;6-7:Baseline,Days 2,4,7,15,29,43,57,85,113,155,183,225;8-9:Baseline,Days 2,4,7,15,29,43,57,85,113,155,183,225,253,281,309,337,365
Population: The pharmacodynamic (PD) analysis set consisted of all dosed participants for whom at least one PD parameter had a baseline value and at least 1 post-baseline measurement available. Participants with data available at each timepoint are presented.
Measure: Mean (Standard Deviation); unit: nmol/L
Groups:
- Cohorts 1-5: Placebo: Participants with screening plasma Lp(a) >=70 nmol/L and <199 nmol/L received placebo matching Olpasiran as a single SC injection on Day 1 in cohorts 1-5.
Arm/Group | Cohorts 1-5: Placebo | Cohort 1: Olpasiran 3 mg | Cohort 2: Olpasiran 9 mg | Cohort 3: Olpasiran 30 mg | Cohort 4 Olpasiran: 75 mg | Cohort 5 Olpasiran: 225 mg | Cohorts 6-9: Placebo | Cohort 6: Olpasiran 9 mg | Cohort 7: Olpasiran 75 mg | Cohort 8: Olpasiran 225 mg | Cohort 9: Olpasiran 675 mg
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 10 | 9 | 9 | 5 | 6
nmol/L
  Change from baseline to Day 2: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 9 | 9 | 9 | 5 | 6
  Change from baseline to Day 2 | 9.740 (11.415) | -17.820 (16.662) | -1.417 (9.409) | 9.412 (13.240) | 1.937 (2.589) | -6.438 (14.001) | -54.862 (91.381) | -4.886 (24.160) | -15.119 (79.070) | -88.586 (105.991) | -86.940 (134.234)
  Change from baseline to Day 4: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 9 | 8 | 8 | 5 | 5
  Change from baseline to Day 4 | 11.450 (13.155) | -13.020 (17.499) | -8.317 (13.271) | 3.862 (12.344) | -23.080 (12.246) | -13.455 (11.489) | -55.527 (100.807) | -33.358 (21.037) | -49.659 (70.520) | -116.986 (71.397) | -146.718 (165.278)
  Change from baseline to Day 7: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 9 | 9 | 9 | 4 | 6
  Change from baseline to Day 7 | 0.410 (12.785) | -24.170 (21.798) | -35.283 (13.307) | -32.272 (7.480) | -45.863 (8.095) | -69.188 (35.265) | -32.389 (99.479) | -77.707 (47.138) | -102.508 (75.135) | -203.215 (112.549) | -204.990 (159.912)
  Change from baseline to Day 15: number analyzed (Participants) | 10 | 6 | 5 | 6 | 6 | 6 | 9 | 9 | 8 | 5 | 6
  Change from baseline to Day 15 | -2.530 (16.293) | -59.137 (28.794) | -76.094 (22.915) | -63.772 (10.074) | -96.580 (11.663) | -98.938 (30.749) | -35.367 (54.976) | -138.618 (38.215) | -208.459 (81.219) | -277.226 (135.590) | -294.890 (176.007)
  Change from baseline to Day 18: number analyzed (Participants) | 10 | 6 | 5 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0
  Change from baseline to Day 18 | -6.940 (15.926) | -71.070 (26.156) | -85.594 (24.516) | -76.222 (13.730) | -108.463 (16.162) | -122.205 (30.732) |  |  |  |  |
  Change from baseline to Day 22: number analyzed (Participants) | 10 | 6 | 5 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0
  Change from baseline to Day 22 | -3.450 (14.989) | -77.853 (25.502) | -93.714 (22.458) | -79.388 (15.566) | -117.813 (19.714) | -126.788 (32.793) |  |  |  |  |
  Change from baseline to Day 29: number analyzed (Participants) | 10 | 6 | 5 | 6 | 6 | 6 | 10 | 9 | 9 | 4 | 5
  Change from baseline to Day 29 | -1.350 (14.355) | -82.037 (26.703) | -104.894 (26.885) | -86.038 (18.938) | -124.713 (23.769) | -134.605 (36.395) | -46.909 (72.951) | -188.740 (37.700) | -270.641 (95.753) | -330.115 (171.096) | -366.214 (199.738)
  Change from baseline to Day 43: number analyzed (Participants) | 10 | 6 | 5 | 6 | 6 | 6 | 8 | 9 | 9 | 4 | 6
  Change from baseline to Day 43 | -7.720 (14.629) | -89.787 (25.866) | -108.734 (28.948) | -90.072 (20.412) | -129.230 (25.491) | -140.572 (36.947) | -33.244 (64.989) | -197.673 (36.630) | -282.841 (95.711) | -257.585 (30.464) | -351.707 (193.404)
  Change from baseline to Day 57: number analyzed (Participants) | 10 | 6 | 5 | 6 | 6 | 6 | 9 | 9 | 9 | 5 | 6
  Change from baseline to Day 57 | 2.620 (11.739) | -87.220 (29.478) | -106.834 (27.834) | -89.955 (20.435) | -129.513 (26.035) | -140.922 (36.663) | -27.973 (104.520) | -200.251 (40.105) | -288.874 (100.724) | -331.386 (166.191) | -353.207 (193.827)
  Change from baseline to Day 71: number analyzed (Participants) | 9 | 6 | 4 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0
  Change from baseline to Day 71 | -0.392 (14.313) | -83.970 (24.076) | -97.518 (24.356) | -88.805 (22.440) | -128.797 (26.709) | -140.572 (37.216) |  |  |  |  |
  Change from baseline to Day 85: number analyzed (Participants) | 9 | 6 | 4 | 6 | 6 | 6 | 9 | 9 | 9 | 5 | 6
  Change from baseline to Day 85 | 2.497 (12.877) | -73.953 (23.337) | -96.318 (23.377) | -85.072 (21.123) | -127.980 (27.181) | -139.255 (36.247) | -35.246 (98.490) | -185.407 (42.933) | -275.519 (95.029) | -330.806 (167.145) | -352.923 (194.316)
  Change from baseline to Day 113: number analyzed (Participants) | 9 | 6 | 4 | 6 | 6 | 6 | 10 | 9 | 9 | 5 | 5
  Change from baseline to Day 113 | 4.697 (6.955) | -63.103 (28.733) | -89.168 (24.019) | -82.338 (24.960) | -123.147 (26.883) | -137.038 (36.491) | -26.599 (83.420) | -162.829 (50.183) | -253.641 (93.836) | -325.526 (168.995) | -276.696 (75.437)
  Change from baseline to Day 155: number analyzed (Participants) | 3 | 0 | 0 | 5 | 5 | 3 | 10 | 9 | 8 | 5 | 5
  Change from baseline to Day 155 | -13.990 (14.136) |  |  | -63.566 (26.356) | -123.076 (29.946) | -144.877 (24.157) | -32.339 (101.724) | -132.696 (52.950) | -195.725 (50.429) | -304.846 (173.370) | -368.258 (212.962)
  Change from baseline to Day 183: number analyzed (Participants) | 2 | 0 | 0 | 0 | 2 | 3 | 10 | 9 | 7 | 5 | 6
  Change from baseline to Day 183 | -20.770 (10.748) |  |  |  | -109.435 (31.304) | -140.143 (25.143) | -32.749 (77.047) | -109.740 (41.868) | -176.781 (51.330) | -291.966 (167.126) | -338.990 (202.609)
  Change from baseline to Day 225: number analyzed (Participants) | 5 | 0 | 0 | 1 | 2 | 5 | 10 | 9 | 9 | 5 | 6
  Change from baseline to Day 225 | -3.902 (18.584) |  |  | -64.100 (NA) — Standard deviation could not be calculated for single participant. | -104.285 (36.607) | -111.892 (27.648) | -15.849 (70.823) | -85.218 (39.572) | -165.297 (89.184) | -257.226 (167.618) | -320.223 (207.672)
  Change from baseline to Day 253: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 4 | 4
  Change from baseline to Day 253 |  |  |  |  |  |  | -101.640 (58.930) |  |  | -276.490 (179.094) | -318.725 (259.063)
  Change from baseline to Day 281: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 5 | 5
  Change from baseline to Day 281 |  |  |  |  |  |  | -96.107 (81.127) |  |  | -230.106 (164.525) | -308.138 (230.671)
  Change from baseline to Day 309: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 5 | 5
  Change from baseline to Day 309 |  |  |  |  |  |  | -117.353 (34.739) |  |  | -215.726 (168.115) | -299.218 (232.143)
  Change from baseline to Day 337: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 4 | 5
  Change from baseline to Day 337 |  |  |  |  |  |  | -113.073 (84.006) |  |  | -198.440 (162.932) | -279.478 (231.897)
  Change from baseline to Day 365: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 5 | 5
  Change from baseline to Day 365 |  |  |  |  |  |  | -81.653 (81.061) |  |  | -170.126 (146.154) | -165.656 (88.637)

6. Secondary Outcome: Percent Change From Baseline in Plasma Lp(a) Levels
Description: Percent change from baseline for plasma Lp(a) by cohort and at scheduled time points during the treatment period were presented.
Time Frame: as for outcome 5
Population: The PD analysis set consisted of all dosed participants for whom at least one PD parameter had a baseline value and at least 1 post-baseline measurement available. Participants with data available at each timepoint are presented.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohorts 1-5: Placebo | Cohort 1: Olpasiran 3 mg | Cohort 2: Olpasiran 9 mg | Cohort 3: Olpasiran 30 mg | Cohort 4 Olpasiran: 75 mg | Cohort 5 Olpasiran: 225 mg | Cohorts 6-9: Placebo | Cohort 6: Olpasiran 9 mg | Cohort 7: Olpasiran 75 mg | Cohort 8: Olpasiran 225 mg | Cohort 9: Olpasiran 675 mg
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 10 | 9 | 9 | 5 | 6
percent change
  Percent change from baseline to Day 2: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 9 | 8 | 9 | 5 | 6
  Percent change from baseline to Day 2 | 8.407 (8.491) | -13.943 (11.951) | -1.094 (7.699) | 8.295 (13.665) | 1.415 (1.925) | -4.027 (9.484) | -13.633 (21.683) | -1.570 (10.443) | -2.088 (20.604) | -21.583 (17.410) | -15.998 (20.674)
  Percent change from baseline to Day 4: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 9 | 8 | 8 | 5 | 5
  Percent change from baseline to Day 4 | 11.483 (13.532) | -9.649 (12.452) | -6.487 (10.577) | 2.462 (12.152) | -17.185 (7.985) | -8.416 (5.613) | -14.608 (23.141) | -12.800 (8.339) | -13.391 (16.046) | -34.553 (16.231) | -30.307 (21.326)
  Percent change from baseline to Day 7: number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 9 | 9 | 9 | 4 | 6
  Percent change from baseline to Day 7 | 0.684 (10.535) | -17.968 (15.135) | -30.135 (14.583) | -34.017 (13.052) | -34.398 (4.843) | -46.725 (15.401) | -7.196 (21.378) | -29.518 (15.778) | -30.979 (14.986) | -58.222 (13.332) | -53.069 (12.226)
  Percent change from baseline to Day 15: number analyzed (Participants) | 10 | 6 | 5 | 6 | 6 | 6 | 9 | 9 | 8 | 5 | 6
  Percent change from baseline to Day 15 | -1.586 (13.188) | -46.805 (17.609) | -61.995 (9.342) | -65.000 (15.685) | -72.512 (5.451) | -69.051 (15.864) | -8.425 (12.997) | -53.145 (15.700) | -66.742 (7.852) | -82.712 (7.795) | -81.166 (5.437)
  Percent change from baseline to Day 18: number analyzed (Participants) | 10 | 6 | 5 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0
  Percent change from baseline to Day 18 | -5.992 (12.779) | -56.826 (15.047) | -69.643 (6.846) | -76.332 (12.228) | -81.178 (6.122) | -84.107 (3.792) |  |  |  |  |
  Percent change from baseline to Day 22: number analyzed (Participants) | 10 | 6 | 5 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0
  Percent change from baseline to Day 22 | -3.064 (11.850) | -62.268 (12.534) | -77.121 (9.413) | -79.157 (11.601) | -87.780 (2.887) | -87.062 (2.254) |  |  |  |  |
  Percent change from baseline to Day 29: number analyzed (Participants) | 10 | 6 | 5 | 6 | 6 | 6 | 10 | 9 | 9 | 4 | 5
  Percent change from baseline to Day 29 | -1.630 (11.948) | -65.771 (14.454) | -85.794 (7.534) | -85.001 (8.595) | -92.577 (1.368) | -92.124 (3.106) | -14.805 (19.160) | -72.210 (15.684) | -85.371 (7.046) | -95.448 (2.665) | -95.872 (1.879)
  Percent change from baseline to Day 43: number analyzed (Participants) | 10 | 6 | 5 | 6 | 6 | 6 | 8 | 9 | 9 | 4 | 6
  Percent change from baseline to Day 43 | -6.503 (11.507) | -72.060 (12.238) | -88.761 (7.479) | -88.558 (6.473) | -95.843 (1.293) | -96.365 (2.122) | -12.075 (21.690) | -75.430 (14.252) | -89.637 (5.632) | -98.226 (0.645) | -98.499 (0.676)
  Percent change from baseline to Day 57: number analyzed (Participants) | 10 | 6 | 5 | 6 | 6 | 6 | 9 | 9 | 9 | 5 | 6
  Percent change from baseline to Day 57 | 1.259 (10.313) | -70.163 (17.697) | -87.421 (9.001) | -88.472 (6.147) | -96.014 (2.073) | -96.685 (1.316) | -4.878 (25.711) | -76.174 (13.755) | -91.230 (6.742) | -98.547 (0.677) | -98.956 (0.400)
  Percent change from baseline to Day 71: number analyzed (Participants) | 9 | 6 | 4 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0
  Percent change from baseline to Day 71 | -1.546 (12.389) | -67.809 (13.524) | -89.962 (4.968) | -86.866 (5.779) | -95.383 (2.145) | -96.332 (1.963) |  |  |  |  |
  Percent change from baseline to Day 85: number analyzed (Participants) | 9 | 6 | 4 | 6 | 6 | 6 | 9 | 9 | 9 | 5 | 6
  Percent change from baseline to Day 85 | 1.275 (11.569) | -59.413 (12.808) | -88.913 (4.425) | -83.628 (8.427) | -94.747 (3.108) | -95.517 (2.334) | -7.875 (20.770) | -70.536 (15.558) | -87.328 (7.434) | -98.275 (0.948) | -98.814 (0.608)
  Percent change from baseline to Day 113: number analyzed (Participants) | 9 | 6 | 4 | 6 | 6 | 6 | 10 | 9 | 9 | 5 | 5
  Percent change from baseline to Day 113 | 3.430 (7.307) | -49.873 (16.496) | -82.051 (7.297) | -79.916 (11.140) | -91.351 (6.866) | -93.926 (2.891) | -6.786 (24.282) | -61.542 (17.396) | -80.484 (11.668) | -96.381 (3.343) | -97.963 (1.142)
  Percent change from baseline to Day 155: number analyzed (Participants) | 3 | 0 | 0 | 5 | 5 | 3 | 10 | 9 | 8 | 5 | 5
  Percent change from baseline to Day 155 | -15.206 (14.391) |  |  | -56.571 (13.156) | -86.424 (11.607) | -88.415 (3.561) | -7.233 (28.936) | -50.331 (20.523) | -68.537 (15.584) | -89.181 (10.167) | -95.757 (4.528)
  Percent change from baseline to Day 183: number analyzed (Participants) | 2 | 0 | 0 | 0 | 2 | 3 | 10 | 9 | 7 | 5 | 6
  Percent change from baseline to Day 183 | -22.300 (6.289) |  |  |  | -76.956 (26.029) | -85.437 (4.356) | -7.884 (23.516) | -41.792 (16.749) | -60.178 (18.037) | -85.355 (11.214) | -93.357 (5.554)
  Percent change from baseline to Day 225: number analyzed (Participants) | 5 | 0 | 0 | 1 | 2 | 5 | 10 | 9 | 9 | 5 | 6
  Percent change from baseline to Day 225 | -4.934 (17.577) |  |  | -84.342 (NA) — Standard deviation could not be calculated for single participant. | -73.464 (29.532) | -81.880 (11.062) | -4.730 (23.419) | -32.228 (14.640) | -51.725 (20.701) | -73.722 (17.160) | -86.702 (12.646)
  Percent change from baseline to Day 253: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 4 | 4
  Percent change from baseline to Day 253 |  |  |  |  |  |  | -24.858 (11.199) |  |  | -76.579 (15.153) | -80.199 (18.262)
  Percent change from baseline to Day 281: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 5 | 5
  Percent change from baseline to Day 281 |  |  |  |  |  |  | -23.787 (22.538) |  |  | -64.718 (19.802) | -75.169 (20.243)
  Percent change from baseline to Day 309: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 5 | 5
  Percent change from baseline to Day 309 |  |  |  |  |  |  | -31.515 (2.142) |  |  | -59.631 (21.986) | -72.336 (19.971)
  Percent change from baseline to Day 337: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 4 | 5
  Percent change from baseline to Day 337 |  |  |  |  |  |  | -26.688 (15.875) |  |  | -52.066 (26.070) | -66.022 (23.528)
  Percent change from baseline to Day 365: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 5 | 5
  Percent change from baseline to Day 365 |  |  |  |  |  |  | -19.333 (15.319) |  |  | -46.309 (23.019) | -56.484 (19.999)

ADVERSE EVENTS:
Time Frame: For all-cause mortality, from randomization until the end of trial completion; median (min, max) time on trial was 8.57 (0.26, 23.95) months. For AE, from first dose of trial drug until the end of trial; median (min, max) duration was 8.54 (0.23, 23.92) months.
Description: All-cause mortality is reported for all participants enrolled/randomized in the trial. Serious AEs and other AEs are reported for all participants who received at least one dose of trial drug.
Arm/Group | Cohorts 1-5: Placebo | Cohorts 6-9: Placebo | Cohort 1: Olpasiran 3 mg | Cohort 2: Olpasiran 9 mg | Cohort 3: Olpasiran 30 mg | Cohort 4 Olpasiran: 75 mg | Cohort 5 Olpasiran: 225 mg | Cohort 6: Olpasiran 9 mg | Cohort 7: Olpasiran 75 mg | Cohort 8: Olpasiran 225 mg | Cohort 9: Olpasiran 675 mg
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/9 | 0/9 | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/9 | 0/9 | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 5/10 | 7/10 | 3/6 | 3/6 | 5/6 | 1/6 | 0/6 | 6/9 | 3/9 | 4/5 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohorts 1-5: Placebo (N=10) | Cohorts 6-9: Placebo (N=10) | Cohort 1: Olpasiran 3 mg (N=6) | Cohort 2: Olpasiran 9 mg (N=6) | Cohort 3: Olpasiran 30 mg (N=6) | Cohort 4 Olpasiran: 75 mg (N=6) | Cohort 5 Olpasiran: 225 mg (N=6) | Cohort 6: Olpasiran 9 mg (N=9) | Cohort 7: Olpasiran 75 mg (N=9) | Cohort 8: Olpasiran 225 mg (N=5) | Cohort 9: Olpasiran 675 mg (N=6)
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac telemetry abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohorts 1-5: Placebo (N=10) | Cohorts 6-9: Placebo (N=10) | Cohort 1: Olpasiran 3 mg (N=6) | Cohort 2: Olpasiran 9 mg (N=6) | Cohort 3: Olpasiran 30 mg (N=6) | Cohort 4 Olpasiran: 75 mg (N=6) | Cohort 5 Olpasiran: 225 mg (N=6) | Cohort 6: Olpasiran 9 mg (N=9) | Cohort 7: Olpasiran 75 mg (N=9) | Cohort 8: Olpasiran 225 mg (N=5) | Cohort 9: Olpasiran 675 mg (N=6)
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Normal tension glaucoma (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Change of bowel habit (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oesophageal spasm (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral mucosal blistering (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Injection site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Medical device site dermatitis (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body tinea (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 2 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Animal scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immunisation reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Smear cervix abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Libido decreased (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pseudofolliculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominoplasty (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mammoplasty (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tenolysis (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diastolic hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/62/NCT03626662/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-08): https://cdn.clinicaltrials.gov/large-docs/62/NCT03626662/SAP_001.pdf